CLINICAL TRIAL: NCT00910624
Title: A Single-Arm Study to Provide Boceprevir Treatment in Subjects With Chronic Hepatitis C Genotype 1 Deemed Nonresponders to Peginterferon/Ribavirin in Previous Schering-Plough Boceprevir Studies
Brief Title: Boceprevir Treatment in Participants With Chronic Hepatitis C Genotype 1 Deemed Nonresponders to Peginterferon/Ribavirin (P05514)
Acronym: PROVIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05514
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BOC + PEG/RBV (Experimental): Participants who enrolled within 2 weeks after the last dose of PEG/RBV in previous protocol received boceprevir (BOC) + peginterferon/ribavirin (PEG/RBV) for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who did not enroll within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
  Interventions: Drug: Boceprevir; Biological: Peginterferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908)

INTERVENTIONS:
Drug: Boceprevir — Boceprevir, 200-mg capsules, 800 mg three times a day (TID) orally (PO)
  Other Names: SCH 503034
Biological: Peginterferon alfa-2b (SCH 54031) — Peginterferon alfa-2b 1.5 µg/kg/week subcutaneously (SC)
  Other Names: PegIntron, PEG
Drug: Ribavirin (SCH 18908) — Ribavirin weight-based dosing (WBD) 600 mg/day to 1400 mg/day PO divided twice daily (BID).
  Other Names: Rebetol, RBV

SUMMARY:
This is a single-arm, multicenter study of boceprevir (BOC) in combination with peginterferon plus ribavirin (PEG/RBV) in adult chronic hepatitis C (CHC) genotype 1 participants who completed their per-protocol defined treatment and did not achieve sustained viral response (SVR) while in the PEG/RBV control arm(s) of an Schering-Plough Research Institute (SPRI) study of BOC combination therapy. Participants who are able to enroll in this study within 2 weeks after the last dose of PEG/RBV in previous protocol are to receive BOC+ PEG/RBV for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who are not able to enroll in this study within 2 weeks after the last dose of PEG/RBV in previous protocol are to receive PEG/RBV for 4 weeks followed by BOC+ PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have been assigned to a PEG/RBV control arm in a previous SPRI study of BOC, must have completed treatment as per protocol, and have been compliant with all study treatment and scheduled procedures within the previous study.
* Participant must have received at least 12 weeks of treatment with PEG/RBV and must have discontinued treatment in the previous study due to the futility rule (as defined in the previous protocol), had virologic breakthrough, or relapse.
* Participant must have had detectable HCV-RNA upon completion of the previous study.
* Participant and participant partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to starting any study treatment and to continue until at least 6 months after the last doses of study drugs, or longer if dictated by local regulations.
* Participant must be willing to give written informed consent.

Exclusion Criteria:

* All participant exclusion criteria from the SPRI clinical study in which the participant participated prior to qualifying for this study will apply in this study, EXCEPT for the following:

  * Treatment with RBV within 90 days and any interferon-alpha within 1 month of the enrollment is not exclusionary in P05514.
  * Participation in any other SPRI clinical trial within 30 days of enrollment in this study is not exclusionary.
  * Use of growth factor at the entry of the study is allowed if it was prescribed in the previous study.
  * Laboratory criteria of thyroid-stimulating hormone (TSH) do not apply. Laboratory criteria of hemoglobin, neutrophils, and platelets do not apply, unless they met dose reduction/interruption/discontinuation criteria in the previous study.
  * Participants who develop moderate depression in the previous study and continue to be stable and well controlled are not excluded
* Participants who had the opportunity to receive boceprevir in the previous study.
* Participants requiring discontinuation, interruption, or dose reduction of RBV for more than 2 weeks in the previous study.
* Participants requiring discontinuation, interruption, or dose reduction of PEG to less than two-thirds of the assigned starting dose for more than 2 weeks in the previous study.
* Participants who experienced a life-threatening SAE considered at least possibly related to study drugs by the investigator or sponsor in the previous study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-06-22 (Actual); Primary Completion 2012-12-07 (Actual); Study Completion 2012-12-07 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Vierling JM, Davis M, Flamm S, Gordon SC, Lawitz E, Yoshida EM, Galati J, Luketic V, McCone J, Jacobson I, Marcellin P, Muir AJ, Poordad F, Pedicone LD, Albrecht J, Brass C, Howe AY, Colvard LY, Helmond FA, Deng W, Treitel M, Wahl J, Bronowicki JP. Boceprevir for chronic HCV genotype 1 infection in patients with prior treatment failure to peginterferon/ribavirin, including prior null response. J Hepatol. 2014 Apr;60(4):748-56. doi: 10.1016/j.jhep.2013.12.013. Epub 2013 Dec 19. PMID 24362076

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 168 participants enrolled and received at least one dose of study medication. Participants were categorized by prior treatment response on the referring study: prior null response, prior partial response, prior relapse, or other.
Groups:
- BOC + PEG/RBV: Prior Null Responders: Participants who achieved "null" response (defined as <2-log10 decrease and detectable HCV RNA at Treatment Week (TW) 12 of PEG/RBV) after completing treatment on the PEG/RBV control arm on a previous SPRI study received BOC + PEG/RBV on the current study for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who were not able to enroll on the current study within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
- BOC + PEG/RBV: Prior Partial Responders: Participants who achieved "partial" response (defined as ≥2-log10 decrease in HCV-RNA by TW 12 and detectable HCV-RNA at end of PEG/RBV) after completing treatment on the PEG/RBV control arm on a previous SPRI study received BOC + PEG/RBV on the current study for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who were not able to enroll on the current study within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
- BOC + PEG/RBV: Prior Relapsers: Participants who achieved "prior relapse" (defined as undetectable HCV-RNA at end of treatment, and detectable HCV-RNA during follow-up period) after completing treatment on the PEG/RBV control arm on a previous SPRI study received BOC + PEG/RBV on the current study for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who were not able to enroll on the current study within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
- BOC + PEG/RBV: Other: Participants who were characterized as "Other" (not in the categories of prior treatment failure as defined by this protocol), after completing treatment on the PEG/RBV control arm on a previous SPRI study, received BOC + PEG/RBV on the current study for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who were not able to enroll on the current study within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
Period: Treatment Phase
Arm/Group | BOC + PEG/RBV: Prior Null Responders | BOC + PEG/RBV: Prior Partial Responders | BOC + PEG/RBV: Prior Relapsers | BOC + PEG/RBV: Other
Started | 52 | 85 | 29 | 2
Completed | 22 | 64 | 20 | 2
Not Completed | 30 | 21 | 9 | 0
Not completed — Adverse Event | 2 | 6 | 6 | 0
Not completed — Treatment Failure | 23 | 10 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Reasons Unrelated To Assigned Treatment | 3 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Non-Compliance With Protocol | 0 | 1 | 1 | 0
Period: Follow-Up Phase
Arm/Group | BOC + PEG/RBV: Prior Null Responders | BOC + PEG/RBV: Prior Partial Responders | BOC + PEG/RBV: Prior Relapsers | BOC + PEG/RBV: Other
Started | 48 | 80 | 29 | 2
Completed | 42 | 76 | 25 | 2
Not Completed | 6 | 4 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 2 | 0
Not completed — Reasons Unrelated To Assigned Treatment | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Withdrew Due To Retreatment Opportunity | 1 | 0 | 0 | 0
Not completed — Administrative | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- BOC + PEG/RBV: Prior Null Responders: Participants who achieved "null" response (defined as <2-log10 decrease and detectable HCV RNA at TW 12 of PEG/RBV) after completing treatment on the PEG/RBV control arm on a previous SPRI study received BOC + PEG/RBV on the current study for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who were not able to enroll on the current study within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
- Total: Total of all reporting groups
Arm/Group | BOC + PEG/RBV: Prior Null Responders | BOC + PEG/RBV: Prior Partial Responders | BOC + PEG/RBV: Prior Relapsers | BOC + PEG/RBV: Other | Total
Number analyzed (Participants) | 52 | 85 | 29 | 2 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (7.7) | 52.6 (8.4) | 53.6 (6.4) | 52.0 (1.4) | 52.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 10 | 1 | 55
  Male | 33 | 60 | 19 | 1 | 113

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at Follow-Up Week 24 (SVR24);
Description: SVR24 was defined as undetectable Hepatitis C Virus ribonucleic acid (HCV-RNA) at Follow-up Week (FW) 24. SVR rates were evaluated by the prior interferon response (e.g., log drop from baseline at TW 4 or TW 12) in the previous studies.
Time Frame: From start of 4-week PEG/RBV lead-in therapy or 44-week BOC/PR treatment through Follow-Up Week (FW) 24 (up to 68 weeks)
Population: All BOC-Treated Participants: All enrolled participants who received at least 1 dose of BOC. Data for 2 "Other" participants were included in the calculations for "BOC + PEG/RBV: All " (n=164). 4 discontinued during the 4-week PEG/RBV lead-in and did not receive BOC and thus were excluded from analysis.
Measure: Number; unit: percentage of participants
Groups:
- BOC + PEG/RBV: All: Participants who enrolled within 2 weeks after the last dose of PEG/RBV in previous SPRI study received boceprevir (BOC) + peginterferon/ribavirin (PEG/RBV) for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who did not enroll within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
Arm/Group | BOC + PEG/RBV: Prior Null Responders | BOC + PEG/RBV: Prior Partial Responders | BOC + PEG/RBV: Prior Relapsers | BOC + PEG/RBV: All
Number analyzed (Participants) | 49 | 85 | 28 | 164
percentage of participants | 41 | 67 | 96 | 65

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Leading to Dose Modification (DM) or Discontinuation (DC), Treatment-Related Serious AEs (SAEs), Neutrophil Count <0.75 × 10^9/L, or Hemoglobin (Hgb) <10 g/dL
Description: AE= any untoward medical occurrence in a participant administered a pharmaceutical product/biologic (at any dose), whether or not considered related to the use of that product. Included the onset of new illness and the exacerbation of pre-existing conditions. Clinically significant laboratory abnormalities that required intervention/additional therapy, required a dose modification, or were associated with a clinical manifestation were considered AEs. SAE= any adverse drug or biologic or device experience occurring at any dose resulting in death, was life-threatening, was persistent or caused significant disability/incapacity, required in-patient hospitalization or prolonged hospitalization, or was a congenital anomaly or birth defect.
Time Frame: From start of 4-week PEG/RBV lead-in therapy or 44-week BOC/PR treatment through FW 24 (up to 68 weeks)
Population: All Treated Participants: All enrolled participants who received at least one dose of treatment.
Measure: Number; unit: percentage of participants
Groups:
- All Treated Participants: Participants who enrolled within 2 weeks after the last dose of PEG/RBV in previous SPRI study received boceprevir (BOC) + peginterferon/ribavirin (PEG/RBV) for up to 44 weeks followed by 24 weeks post-treatment follow-up. Participants who did not enroll within 2 weeks after the last dose of PEG/RBV in previous protocol received PEG/RBV for 4 weeks followed by BOC + PEG/RBV for up to 44 weeks, with 24 weeks post-treatment follow-up.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 168
percentage of participants
  AEs Leading to DC | 8
  AEs Leading to DM | 35
  All Treatment-Related SAEs | 7
  SAEs Related to BOC+PEG or BOC+P/R | 4
  Neutrophil Count <0.75 × 10^9/L | 25
  Hgb <10 g/dL | 53

3. Secondary Outcome: Percentage of Participants With Early Virologic Response (EVR)
Description: EVR was defined as undetectable HCV-RNA at TW 12 of BOC + PEG/RBV. EVR rates were evaluated by the prior interferon response (e.g., log drop from baseline at TW 4 or TW 12) in the previous studies.
Time Frame: From TW 1 to TW 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | BOC + PEG/RBV: Prior Null Responders | BOC + PEG/RBV: Prior Partial Responders | BOC + PEG/RBV: Prior Relapsers | BOC + PEG/RBV: All
Number analyzed (Participants) | 49 | 85 | 28 | 164
percentage of participants | 49 | 76 | 100 | 73

ADVERSE EVENTS:
Time Frame: From start of 4-week PEG/RBV lead-in therapy or 44-week BOC/PR treatment through FW 24 (up to 68 weeks)
Description: Only treatment-emergent AEs occurring on the present study (NCT00910624) and AEs occurring during the follow-up period of the present study are reported.
Arm/Group | All Treated Participants
Serious Adverse Events (participants affected / at risk) | 18/168
Other Adverse Events (participants affected / at risk) | 161/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Participants (N=168)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Injection site abscess (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Participants (N=168)
Anaemia (Blood and lymphatic system disorders) | 83 (141)
Leukopenia (Blood and lymphatic system disorders) | 15 (19)
Neutropenia (Blood and lymphatic system disorders) | 38 (53)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (15)
Abdominal pain (Gastrointestinal disorders) | 12 (16)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 37 (49)
Dry mouth (Gastrointestinal disorders) | 10 (11)
Dysgeusia (Gastrointestinal disorders) | 59 (64)
Dyspepsia (Gastrointestinal disorders) | 12 (12)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (13)
Nausea (Gastrointestinal disorders) | 52 (59)
Vomiting (Gastrointestinal disorders) | 14 (16)
Asthenia (General disorders) | 23 (27)
Chills (General disorders) | 27 (28)
Fatigue (General disorders) | 81 (104)
Influenza like illness (General disorders) | 35 (37)
Injection site reaction (General disorders) | 16 (16)
Irritability (General disorders) | 25 (32)
Pain (General disorders) | 10 (12)
Pyrexia (General disorders) | 22 (27)
Weight decreased (Investigations) | 15 (18)
Decreased appetite (Metabolism and nutrition disorders) | 35 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (18)
Disturbance in attention (Nervous system disorders) | 11 (11)
Dizziness (Nervous system disorders) | 27 (32)
Headache (Nervous system disorders) | 45 (50)
Depression (Psychiatric disorders) | 22 (25)
Insomnia (Psychiatric disorders) | 40 (52)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (30)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (35)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (29)
Dry skin (Skin and subcutaneous tissue disorders) | 28 (31)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (25)
Rash (Skin and subcutaneous tissue disorders) | 24 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor, and further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.